CLINICAL TRIAL: NCT02925546
Title: An Open Label, Randomized, Single Dose, Crossover Study to Determine the Pharmacokinetics of Three Tablet Formulations of GSK2798745 in Healthy Subjects
Brief Title: A Phase I Study to Assess the Pharmacokinetics of GSK2798745 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204725
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure, Congestive
Keywords: Healthy; Pharmacokinetics; Phase I; GSK2798745; Tablet
MeSH Terms: conditions — Heart Failure | interventions — long-chain-aldehyde dehydrogenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK2798745 ABCD treatment sequence (Experimental): Subjects will be given 2.4 mg single oral doses of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)
- GSK2798745 CABD treatment sequence (Experimental): Subjects will be given 2.4 mg GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), 2.4 mg single oral doses of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)
- GSK2798745 ACBD treatment sequence (Experimental): Subjects will be given 2.4 mg single oral doses of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), 2.4 mg GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)
- GSK2798745 BACD treatment sequence (Experimental): Subjects will be given 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), 2.4 mg of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), 2.4 mg GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)
- GSK2798745 BCAD treatment sequence (Experimental): Subjects will be given 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), 2.4 mg GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), 2.4 mg single oral doses of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)
- GSK2798745 CBAD treatment sequence (Experimental): Subjects will be given 2.4 mg GSK2798745 (milled API with SLS and hypromellose) in fasted state (treatment C), 2.4 mg of GSK2798745 (micronized API with SLS and hypromellose) in fasted state (treatment B), 2.4 mg single oral doses of GSK2798745 (micronized API without SLS and hypromellose) in fasted state (treatment A), and GSK2798745 tablet in fed state (treatment D) in either treatment periods 1, 2, or 3; the three treatment periods will each be separated by a minimum washout period of 7 days
  Interventions: Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A); Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B); Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C)

INTERVENTIONS:
Drug: GSK2798745 Micronized API without SLS and hypermellose (Tablet A) — This is an immediate release tablet containing 2.4 mg of micronized GSK2798745 API; to be administered orally with 240 mL of water under fasted/fed conditions
Drug: GSK2798745 Micronized API with SLS and hypermellose (Tablet B) — This is an immediate release tablet containing 2.4 mg of micronized GSK2798745 API with SLS and hypermellose; to be administered orally in fasted/fed conditions with 240 mL of water
Drug: GSK2798745 milled API without SLS and hypermellose (Tablet C) — This is an immediate release tablet containing 2.4 mg of milled GSK2798745 API with SLS and hypermellose; to be administered orally in fasted/fed conditions, with 240 mL of water

SUMMARY:
GSK2798745 is being developed as a novel therapeutic intervention for the treatment of pulmonary edema associated with heart failure (HF) and is currently under investigation in the form of a compounded capsule. This is an open-label, randomized, single-dose, crossover study with the purpose to determine the pharmacokinetics (PK) of three 2.4 milligrams (mg) tablet formulations of GSK2798745 in 12 healthy subjects. The three formulations developed for this study will be micronized GSK2798745 active pharmaceutical ingredient (API) (Tablet A), micronized GSK2798745 API with sodium lauryl sulfate (SLS) and hypromellose (Tablet B), milled GSK2798745 API with SLS and hypermellose (Tablet C), and Tablet D, which will be either A/B/C based on interim PK analysis of data from the first three treatment periods.

Following a 30-day screening period, subjects will be randomized to one of the 6 treatment sequences: Treatment sequence 1: ABCD, 2=CABD, 3=ACBD, 4=BACD, 5=BCAD, 6=CBAD over three 4-day treatment periods. For treatment period 4, the best formulation based on the interim analysis data from the three treatment periods will be evaluated under fed conditions. Each treatment period will be separated by a minimum of 7 (+14)-day washout period. The total duration of participation in the study will be approximately 11 weeks including the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Body weight >=50 kg and body mass index within the range 18 - 32 kilogram (kg)/meter (m)^2 (inclusive)
* Male or female of non-child bearing potential:

A male subject with a female partner of child bearing potential is eligible to participate if he agrees to use contraception as mentioned in the protocol during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period A female subject is eligible to participate if she is not a woman of childbearing potential (WOCBP) as defined in the protocol.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol

Exclusion Criteria:

* History of acute coronary syndromes including unstable angina or myocardial infarction within 6 months of screening
* History of stroke or seizure disorder within 5 years of Screening
* Active ulcer disease or gastrointestinal bleeding at the time of screening
* Alanine transaminase (ALT) and bilirubin >1.5x Upper limit of normal (ULN) is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QT interval corrected according to Fridericia's formula (QTcF) >450 milliseconds (msec)
* History or current evidence of any serious or clinically significant gastrointestinal, renal, endocrine, neurologic, hematologic or other condition that is uncontrolled on permitted therapies or that would, in the opinion of the investigator or the Medical Monitor, make the subject unsuitable for inclusion in this study
* Urinary cotinine levels indicative of current smoking or regular use of tobacco- or nicotine-containing products at time of screening (cotinine levels >200 nanogram [ng]/millimeter [mL])
* History of alcohol abuse within 6 months of the study based on the following criteria:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits

* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen, positive hepatitis C antibody test result at screening or within 3 months of screening.
* A positive test for human immunodeficiency virus antibody
* A positive pre-study drug/alcohol screen
* A screening cardiac Troponin level > ULN
* Use of another investigational product in a clinical study within the following time period prior to the first administration of study medication in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first administration of study medication.
* Unable to refrain from the use of prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) except permitted medications listed in the protocol, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and/ or sponsor the medication will not interfere with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of GSK2798745 | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in each of the treatment periods
  AUC will be determined following a single oral dose of GSK2798745 under fasted conditions (Treatment periods 1-3) and fed conditions (Treatment period 4)
Maximum plasma concentration (Cmax) of GSK2798745 | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in each of the treatment periods
  Cmax will be determined following a single oral dose of GSK2798745 under fasted conditions (Treatment periods 1-3) and fed conditions (Treatment period 4)

SECONDARY OUTCOMES:
Time to maximum observed concentration (Tmax) of GSK2798745 | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in each of the treatment periods
  Tmax will be determined following a single oral dose of GSK2798745
Elimination half-life (T1/2) of GSK2798745 | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in each of the treatment periods
  T1/2 will be determined following a single oral dose of GSK2798745
AUC of GSK2798745 following a standard Food Drug Administration (FDA) high fat, high calorie meal | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in treatment period 4
  The effect of food on the PK of one of the three tablet formulations of GSK2798745 will be assessed by AUC following a single oral dose of GSK2798745 which was admininstered 30 minutes after start of a FDA high fat, high-calorie meal
Cmax of GSK2798745 following a standard FDA high fat, high calorie meal | Blood samples will be collected at the following time points: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 15 (Day 1), 24 and 36 (Day 2), 48 (Day 3) and 72 hours (Day 4) post dose in treatment period 4
  The effect of food on the pharmacokinetics of one of the three tablet formulations of GSK2798745 will be assessed by Cmax following a single oral dose of GSK2798745 which was admininstered 30 minutes after start of a FDA high fat, high-calorie meal
Systolic and diastolic blood pressure as a measure of safety and tolerability of GSK2798745 | Up to 11 weeks
  This will be measured in triplicate in a semi-supine position after 5 minutes rest
Pulse rate as a measure of safety and tolerability of GSK2798745 | Up to 11 weeks
  This will be measured in triplicate in a semi-supine position after 5 minutes rest
Respiratory rate as a measure of safety and tolerability of GSK2798745 | Up to 11 weeks
  This will be measured in triplicate in a semi-supine position after 5 minutes rest
Safety and tolerability of single dose of GSK2798745 as assessed by electorcardiograms (ECGs) | Up to 11 weeks
  Triplicate twelve-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected according to Fridericia's formula (QTcF) intervals. ECGs will be measured after resting in semi-supine position for 5 minutes
Safety and tolerability of single dose of GSK2798745 as assessed by hematology | At Baseline (Day -1)
  Hematology parameters include platelet, red blood cell counts, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils, and basophils
Safety and tolerability of single dose of GSK2798745 as assessed by clinical chemistry | At Baseline (Day -1)
  Clinical chemistry parameters included Blood urea nitrogen, Creatinine, Glucose (fasting), Uric acid, Potassium, Sodium, Calcium, Chloride, Total Protein, Albumin, and creatine phosphokinase
Safety and tolerability of single dose of GSK2798745 as assessed by urinalysis | At Baseline (Day -1)
  The following urinalysis parameters will be measured: Protein, Blood, Ketones, glucose, specific gravity, power of hydrogen (pH) by dipstick method. If blood or protein is abnormal, microscopic examination will be performed
Safety and tolerability of single dose of GSK2798745 as assessed by liver function tests (LFTs) | At Baseline (Day -1)
  The following parameters will be measured: Aspartate aminotransferase, Alanine aminotransferase, Alkaline phosphatase, Total and direct bilirubin
Safety and tolerability of single dose of GSK2798745 as assessed by weight assessments | Up to 11 weeks
Safety and tolerability of single dose of GSK2798745 as assessed by appetite assessments | Up to 11 weeks
  Subject will be administered a four-item Simplified Nutritional Assessment Questionnaire (SNAQ) on Days -1 and 2 of each treatment period and at the Follow Up Visit; the sum of the scores for the individual items will constitute the SNAQ
Safety and tolerability of single dose of GSK2798745 as assessed by troponin measurement | At Baseline (Day -1) and 24 hours post dose on Day 2
Number of subjects with any adverse events (AEs) as a measure of safety and tolerability of GSK2798745 | Up to 11 weeks
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States